CLINICAL TRIAL: NCT02430272
Title: Anticholinergic Premedication Induced Fever in Pediatric Ambulatory Anesthesia With Ketamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Won Joo Choe, M.D., Ph.D., Associate professor,, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DSC-01-choe
Record Dates: First submitted 2015-04-22; First posted 2015-04-30 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Fever
Keywords: Child; outpatient; premedication
MeSH Terms: conditions — Fever | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Anticholinergic premedication (Experimental): Premedication with 0.005mg/Kg of glycopyrrolate
  Interventions: Drug: Glycopyrrolate
- Control group (No Intervention): Same volume of normal saline

INTERVENTIONS:
Drug: Glycopyrrolate — Intravenously administered 0.005mg/Kg of glycopyrrolate in intervention group
  Arms: Anticholinergic premedication

SUMMARY:
Anticholinergic drugs have traditionally been used for their antisialagogue properties. But use of anticholinergic drugs can interfere with thermoregulation via inhibition of the parasympathetically mediated sweat secretion. Sweating inhibition can reduce heat elimination, and children's thermoregulation depend more on sweating than adults and they can become hyperthermic when given these agents.

The investigators evaluated the fever-causing effects of adjunctive anticholinergics in children under general anesthesia using ketamine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status classification I
* underwent surgery between 8 to 9 am
* undergoing ambulatory anesthesia with ketamine

Exclusion Criteria:

* who required endotracheal intubation
* who were administered with medications other than ketamine

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body temperature | every 30 minutes from base line ( up to 90min )
  measured body temperature at three times in both ears and the highest value was selected.

SECONDARY OUTCOMES:
Oral secretion (VAS) | up to operative end
  Oral secretion during the whole procedure was recorded by the researcher

CONTACTS AND LOCATIONS:
Overall Officials: Won Joo Choe, M.D. Ph.D, Study Chair — Inje Univ.
Locations (1):
- Ilsan Paik hospital, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim KW, Choe WJ, Kim JH, Kim KT, Lee SI, Park JS, Kim JW, Heo MH. Anticholinergic premedication-induced fever in paediatric ambulatory ketamine anaesthesia. J Int Med Res. 2016 Aug;44(4):817-23. doi: 10.1177/0300060515595649. Epub 2016 May 25. PMID 27225859